CLINICAL TRIAL: NCT01858064
Title: Predicting Treatment Response to Stimulants in Adult ADHD Using Functional Magnetic Resonance Imaging
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Competing Departmental Studies
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013000956
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: ADHD
Keywords: ADHD; OROS-MPH; Adults; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OROS-MPH (Experimental): OROS-MPH is administered in capsule form daily, beginning at 36 mg/day and titrated on a weekly basis for 3 weeks in increments of 18-36 mg/day to a maximum daily dose of 90mg/day.
  Interventions: Drug: OROS-MPH

INTERVENTIONS:
Drug: OROS-MPH — Capsule administered daily, beginning at 36 mg/day and titrated on a weekly basis for 3 weeks in increments of 18-36 mg/day to a maximum daily dose of 90 mg/day.

SUMMARY:
The primary aim of this study is to assess the predictability of treatment response to stimulants in adults with ADHD using functional magnetic resonance

This study will be a six-week, open-label study including adults ranging from age 18-55 with ADHD.

DETAILED DESCRIPTION:
Certain brain characteristics have been identified in individuals with persistent and remitted ADHD. We predict that neural functional connectivity; specifically decreases in connectivity between the posterior cingulated cortex and medial prefrontal cortex, as well as decreases in anticorrelations between the medial prefrontal cortex and dorsolateral prefrontal cortex, will predict greater response to stimulant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 18-55 years
* Right handed
* A diagnosis current of childhood onset ADHD, according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) based on clinical assessment
* A score of > 20 on the Adult ADHD Investigator Symptom Report Scale (AISRS) or a CGI-Severity score of > 4 (moderate severity)

Exclusion Criteria:

* A history of non-response or intolerance to stimulants at adequate doses as determined by the clinician
* Pregnant or nursing females
* Serious, unstable medical illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinologic (thyroid), neurologic (seizure), immunologic, or hematologic disease
* Glaucoma
* Clinically unstable psychiatric conditions including suicidality, homocidality, bipolar disorder, psychosis, or lifetime history of a clinically serious condition potentially exacerbated by a stimulant, such as mania or psychosis
* Tics or diagnosis of Tourette's syndrome
* Current (within 3 months) DSM-IV criteria for abuse or dependence with any psychoactive substance other than nicotine
* Current use of psychotropic medications
* Current use of MAO Inhibitor or use within the past two weeks
* Claustrophobia or an standard contraindications to MRI scanning (metal in body)
* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent or grandchild

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Adult Investigator Rating Scale | Baseline to 6 weeks
  AISRS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States